CLINICAL TRIAL: NCT01030848
Title: Time-dependent Improvement of Functional Outcome Following LCS Rotating Platform TKR - A Prospective Longitudinal Study With Repetitive Measures of KOOS
Brief Title: Time-dependent Improvement of Functional Outcome Following LCS Rotating Platform TKR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Tor Kjetil Nerhus/ Consultant orthopaedic surgeon, Martina Hansens Hospital
Other Study IDs: TKN-001; 19039 (NSD) (Registry Identifier: Norwegian Privacy Ombudsman for Research)
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Osteoarthritis; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with knee osteoarthritis
  Interventions: Device: Total Knee Replacement (LCS rotating platform)

INTERVENTIONS:
Device: Total Knee Replacement (LCS rotating platform)

SUMMARY:
The objective of this prospective study is to determine (1) the time course of patient-relevant functional outcome evaluated by the Knee injury and Osteoarthritis Outcome Score (KOOS) and (2) the time course of range of motion (ROM) the first four years following TKR using the LCS rotating platform prosthesis. Improvement of patient self-reported pain and daily function during the study period, are of particular interest.

ELIGIBILITY:
Inclusion Criteria:

* patients with knee osteoarthritis
* admitted for total knee replacement
* no rheumatoid arthritis
* no previous knee infection
* age 40-85 years

Exclusion Criteria:

-

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients operated with total knee arthroplasty at Martina Hansens Hospital
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2003-02; Primary Completion 2007-09 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score | Preoperative and 6 weeks, 3 months, 6 months, 1 year, 2 years and 4 years postoperatively

SECONDARY OUTCOMES:
Range of Motion (ROM) | Preoperative and 6 weeks, 3 months, 6 months, 1 year, 2 years and 4 years postoperatively
Knee injury and Osteoarthritis Outcome Score | 10 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Tor Kjetil Nerhus, MD, Principal Investigator — Martina Hansens Hospital
Locations (1):
- Martina Hansens Hospital, Bærum, Bærum, Norway